CLINICAL TRIAL: NCT04996355
Title: Prospective Observation on the Accuracy of in Vitro Screening of Colorectal Cancer Chemotherapy Drugs Based on Organoids-on-a-chip
Brief Title: Organoids-on-a-chip for Colorectal Cancer and in Vitro Screening of Chemotherapeutic Drugs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PHB148-001
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Neoplasms; Organoids
Keywords: organoids; colorectal cancer; drug screening; organoids-on-a-chip
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue，blood sample,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: comprehensive treatment after MDT discussion — The comprehensive treatment plan was determined through MDT discussion, which was completed by the Department of Gastrointestinal Surgery, Peking University People's Hospital.
  The following regimens will be tested with organoids-on-a-chip：
  1. 5-FU
  2. Oxaliplatin
  3. Irinotecan
  4. 5-FU+ Oxaliplatin
  5. 5-FU+ Irinotecan
  6. 5-FU+ Oxaliplatin+ Irinotecan
  7. 5-FU+Cetuximab
  8. Cetuximab
  9. Regorafenib

SUMMARY:
The individualized treatment of tumors has always been an urgent problem in clinical practice. Organoids-on-a-chip can reflect the heterogeneity of tumors and is a good model for in vitro anticancer drug screening. In this study, surgical specimens of patients with advanced colorectal cancer will be collected for organoid culture and organoids-on-a- chip. Use organoids-on-a-chip to screen tumor chemotherapy drugs, compare the results of patients' actual medication regimens, and study the guiding role of organoids in the formulation of precise tumor treatment plans. The investigators will compare the response of organoids to drugs in vitro with the patient's response to actual chemotherapy and targeted drugs and explore the feasibility and accuracy of organoids-on-a-chip based drug screening for advanced colorectal cancer. The project will establish a screening platform for chemotherapeutic drugs and targeted drugs based on colorectal cancer organoids to quickly and accurately formulate personalized treatment plans for clinical patients.

DETAILED DESCRIPTION:
1. Establish and identify colorectal cancer organoid chip culture system: collect tumor tissues and normal tissues from patients with advanced colorectal cancer. Culture primary organoids, and organoids derived from normal mucosal tissues as controls. Validate tumor organoids and organoid chips by morphology (HE, immunohistochemical staining) and gene sequencing (target-seq) methods.
2. After each enrolled patient undergoes MDT discussion, chemotherapy is given to the patient according to the existing clinical guidelines and clinical pathways for colorectal cancer. Meanwhile, in vitro drug screening based on colorectal cancer organoid chips is conducted. Collect target gene sequencing results and common clinical medication plans. Local recurrence rate, disease progression-free survival rate and overall survival rate will be followed up for 2 years.
3. Compare the patient's response to the actual medication regimen and organoids in vitro drug screening based on organoids-on-a-chip, and evaluate the accuracy, specificity and sensitivity of organoids-on-a-chip for in vitro drug screening.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate the study and sign informed consent, with good compliance and follow-up;
2. Patients who can tolerate chemotherapy and targeted therapy, ECOG≤1 point;
3. Patients with advanced colorectal cancer diagnosed by pathology and imaging; 4. Neutrophil count ≥2.0×10^9/L, Platelet count ≥100×10^9/L, Hemoglobin ≥90g/L, Serum total bilirubin ≤ 1.5 times the upper limit of normal value, Alanine aminotransferase and Aspartate aminotransferase ≤ 1.5 times the upper limit of normal value, and Serum creatinine ≤ 1.5 times the upper limit of normal value.

Exclusion Criteria:

1. Patients who cannot obtain enough tissue for gene test and the organoids-on-a-chip culture;
2. Patients previously combined with other malignant tumors of other organs;
3. Patients who need emergency operation due to perforation and obstruction；
4. Patients who have active hepatitis, HIV (+) and other conditions that cannot tolerate chemotherapy;
5. Patients who have serious heart and lung diseases, vascular diseases, mental diseases or drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each patient should complete the following items within two weeks of admission, which should be completed by the Gastrointestinal Surgery Department of Peking University People's Hospital:
  1. Complete medical history；
  2. Detailed personal data；
  3. Current treatment；
  4. Physical examination；
  5. Blood routine examination；
  6. Liver and kidney function examination；
  7. Tumor marker examination included CEA, CA199, CA724, AFP；
  8. Infection, blood coagulation examination；
  9. ECG, Ultrasound, Chest radiograph, Gastroenterostomy, and Imaging examination of tumor lesions.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy, specificity and sensitivity of organoids-on-chip for drug sreening | 2 years
  The accuracy, specificity and sensitivity of in vitro drug sensitivity screening based on organoid-chips to predict the effect of chemotherapy (traditional chemotherapy, targeted therapy) for advanced colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Yingjiang Ye, PHD&MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China